CLINICAL TRIAL: NCT01621815
Title: Variance of Video Games Playing Patterns Among Adolescents With Psychiatric Disorders: Diagnostical and Dynamic Meanings
Brief Title: Variance of Video Games Playing Patterns Among Adolescents With Psychiatric Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shalvata Mental Health Center (Other)
Responsible Party: Principal Investigator, Aviv Segev, Principal Investigator, Shalvata Mental Health Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: SH-12-13
Record Dates: First submitted 2012-06-14; First posted 2012-06-18 (Estimated); Last update posted 2015-05-20 (Estimated); Status verified 2015-05

CONDITIONS: ADHD; Conduct; Depression; Anxiety; PDD
Keywords: ADHD; Attention Deficit/Hyperactivity Disorder; Conduct; Depression; Anxiety; PDD; Pervasive Developmental Disorders
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Behavior; Depression; Anxiety Disorders; Child Development Disorders, Pervasive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Anxiety and Depression (Active Comparator): Adolescents diagnosed with anxiety and/or depression
  Interventions: Behavioral: Video Game
- ADD (Active Comparator): Adolescents diagnosed with ADD (without hyperactive element)
  Interventions: Behavioral: Video Game
- ADHD, Behavioral (Active Comparator): Adolescents diagnosed with ADHD (with hyperactivity), with or without behavioral problems
  Interventions: Behavioral: Video Game
- PDD (Active Comparator): Adolescents diagnosed with PDD Spectrum Disorders
  Interventions: Behavioral: Video Game
- Control (Active Comparator): Adolescents without a psychiatric diagnosis
  Interventions: Behavioral: Video Game

INTERVENTIONS:
Behavioral: Video Game — Playing various video games: RPG, Race, FPS, Strategy
  Other Names: Video Games; Computer Games; RPG; Role Playing Games; FPS; First Person Shooter; Strategy

SUMMARY:
As the use of video games (VG) is rapidly increasing, many studies have tries to understand the effects of VG on the children and adolescents playing them.

Most of the research was directed towards negative effects (especially violence, attention and school performance), producing mixed results.

Recently, more studies had focused their attention on the opposite angle: The influence of the player's mental and behavioral parameters, influencing his VG playing patterns. The focus of most of these researches was time of playing, addictive patterns and exposure to violence.

The current study will try to characterize the variance of VG playing pattern among adolescents diagnosed with psychiatric disorders, in order to better under the rich interaction between a player and his VG, and to understand whether VG playing patterns holds diagnostical clues for the child's diagnosis and his inner world.

DETAILED DESCRIPTION:
The participants will be asked to attend 2 session, 2 hours each, at 3-14 days interval.

At the first session, after signing consent form, will asked to fill out questionaires regarding demographic data, personality, empathy trait, aggression state and trait and computer games usage.

also, they will be asked to complete HTP and TAT psycho-diagnostic tests. Then, using heart rate variability (HRV) and Galvanic skin response (GSR), monitor of sympathetic tonus will be measured while playing a shooting and race game.

At the end of the first session, they will be asked to fill additional aggression state questionaire.

On the second session, monitored by HRV and GSR, they will be asked to play a role playing game (RPG) and real-time strategy game (RTS). At the end of session, they will be asked to fill additional aggression state questionaire.

Parameters of playing patterns collected from the VG will be recorded and analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Age 13-18
* Diagnosis matching one of the defined research arms, made by a childhood and adolescents psychiatry specialist
* Playing various computer games regularly, for at least 2 years
* Informed consent has been given by the minor and his parents

Exclusion Criteria:

* Organic sensory depravation (blindness, deafness)
* Motor dysfunction, relevant of using keyboard, mouse or remote
* Additional psychiatric diagnosis, apart the one matching the arm to which he was allocated
* Using illicit drugs during the previous 48 hours

Ages: 13 Years to 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 46 (Actual)
Dates: Start 2012-07; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aviv Segev, MD, Principal Investigator — Shalvata MHC
Locations (1):
- Shalvata MHC, Hod HaSharon, Israel